CLINICAL TRIAL: NCT00972257
Title: Quality of 24-hour Intraocular Pressure Control Obtained With Dorzolamide/Timolol Fixed Combination (DTFC) Compared With the Brimonidine/Timolol Fixed Combination (BTFC) in Subjects With Primary Open-angle Glaucoma
Brief Title: 24-hr Intraocular Pressure Control With Dorzolamide/Timolol vs the Brimonidine/Timolol Fixed Combination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A5132
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
Keywords: 24-hour IOP control; primary open-angle glaucoma; brimonidine/timolol; dorzolamide/timolol
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle | interventions — Therapeutics; dorzolamide; Timolol; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: Dorzolamide/Timolol (Active Comparator)
  Interventions: Drug: treatment with dorzolamide/timolol
- Treatment with Brimonidine/Timolol (Active Comparator)
  Interventions: Drug: treatment with brimonidine/timolol

INTERVENTIONS:
Drug: treatment with dorzolamide/timolol — 24-hour IOP control with the two fixed combinations
  Arms: Drug: Dorzolamide/Timolol
Drug: treatment with brimonidine/timolol — 24-hour pressure control with brimonidine/timolol
  Arms: Treatment with Brimonidine/Timolol

SUMMARY:
The proposed study will compare for the first time the quality of 24-hour IOP control with Brimonidine/Timolol fixed combination (BTFC) versus Dorzolamide/Timolol fixed combination (DTFC) after a run-in period of 2 months with timolol. This crossover comparison may determine the real efficacy of the two fixed combinations and the design of the proposed study may explain for the first time why the 24-hour IOP reduction provided by BTFC is less than might be anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive, newly diagnosed or previously untreated POAG patients
* Patients with typical glaucomatous disc, or visual field damage
* Patient must have IOP (at 10:00 ± 1 hour)greater than 25 mm Hg

Exclusion Criteria:

* Uncontrolled glaucoma
* Distance best corrected Snellen visual acuity worse than 1/10
* Contraindications to brimonidine or dorzolamide and β-blockers
* History of lack of response (<10% morning IOP reduction) to any medication
* Patient can not understand the instructions and adhere to medications
* Patient is a female of childbearing potential or lactating mother
* Prior surgery, past use of steroids (within 2 months)
* Severe dry eyes and use of contact lenses
* History of non-adherence
* Patients with closed angles

Ages: 29 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To compare the quality of 24-hour IOP control after 2 months of chronic therapy with the Dorzolamide/Timolol fixed combination versus the Brimonidine/Timolol fixed combination in primary open-angle glaucoma. | 3 months

SECONDARY OUTCOMES:
Assess fluctuation of 24-hour pressure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Konstas, MD, phD, Principal Investigator — Head of Glaucoma Unit
Locations (1):
- Glaucoma Unit, 1st University Dept of Ophthalmology, Thessaloniki, Greece

REFERENCES:
- [Derived] Konstas AG, Quaranta L, Yan DB, Mikropoulos DG, Riva I, Gill NK, Barton K, Haidich AB. Twenty-four hour efficacy with the dorzolamide/timolol-fixed combination compared with the brimonidine/timolol-fixed combination in primary open-angle glaucoma. Eye (Lond). 2012 Jan;26(1):80-7. doi: 10.1038/eye.2011.239. Epub 2011 Sep 30. PMID 21960068